CLINICAL TRIAL: NCT02589769
Title: Effects of Reduction in Saturated Fat on Cholesterol and Lipoproteins in Lean and Obese Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tine Mejlbo Sundfør, M.Sc in Nutrition, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1786 (REK(
Record Dates: First submitted 2015-06-16; First posted 2015-10-28 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-09

CONDITIONS: Cardiovascular Disease; Dietary Modification; Cardiovascular Risk Factors
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fats, Unsaturated; Fatty Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- unsaturated fat (Experimental): an intervention diet substituting unsaturated fats from oil and nuts for saturated fats from meat and dairy foods
  Interventions: Other: unsaturated fat for saturated fat
- saturated fat (Active Comparator): a control diet with whole fat dairy and meat with saturated fats that are not fat reduced.
  Interventions: Other: saturated fat

INTERVENTIONS:
Other: unsaturated fat for saturated fat — Substituting unsaturated fat for saturated fat
  Arms: unsaturated fat
Other: saturated fat — a control diet with whole fat dairy and meat with saturated fats that are not fat reduced
  Arms: saturated fat

SUMMARY:
A randomized controlled clinical trial comparing the effect of substitution of unsaturated fat from nuts and oils for saturated fat from meat and dairy foods on serum lipids in normal weight and obese subjects with elevated LDL cholesterol.

DETAILED DESCRIPTION:
Background: Increased intake of saturated fat may influence LDL cholesterol and other cardiovascular risk factors different in normal weight and obese subjects. Methods: The study is a randomized controlled clinical trial in 84 men and women between 21 to 70 years with normal BMI (25 kg/m2) or obesity (BMI 30-45 kg/m2) and elevated LDL cholesterol (>3.0 mmol/l). Dietary intervention: Randomization will be to one of two balanced weight maintenance Mediterranean-type diets that differ in their fat sources: an intervention diet substituting unsaturated fats from oil and nuts for saturated fats from meat and dairy foods, and a control diet with whole fat dairy and meat with saturated fats that are not fat reduced.

Primary research question: Compare the effect of substitution of unsaturated fat from nuts and oils for saturated fat from meat and dairy foods on serum lipids in normal weight and obese subjects with elevated LDL cholesterol.

Secondary research questions: Compare the effect of substitution of unsaturated fat from nuts and oils for saturated fat on cardiometabolic risk factors including insulin resistance, inflammation and serum PCSK9 in normal weight and obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 21 to 70 years with normal BMI (25 kg/m2) or obesity (BMI 30-45 kg/m2) and elevated LDL cholesterol (> 3.0 mmol/l).

Exclusion Criteria:

* Diabetes types 1 and 2
* History of CVD including myocardial infarction, percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG), stroke, transient ischemic attack (TIA) or other atherosclerotic disease, eating disorder and other secondary causes of hyperlipidemia.
* Use of statins or other cholesterol-modifying drugs.
* Genetic lipid disorder.
* Gastrointestinal disorders that limit food choices.
* Psychiatric illness, drug or alcohol abuse.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-09; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Serum lipids in normal weight and obese subjects with elevated LDL cholesterol. | 10 weeks
  Compare the effect of substitution of unsaturated fat from nuts and oils for saturated fat from meat and dairy foods on serum lipids in normal weight and obese subjects with elevated LDL cholesterol.

SECONDARY OUTCOMES:
C-reactive protein in normal weight and obese individuals | 10 weeks
  Compare the effect of substitution of unsaturated fat from nuts and oils for saturated fat on c-reactive protein in normal weight and obese individuals
Serum PCSK9 in normal weight and obese individuals | 10 weeks
  Compare the effect of substitution of unsaturated fat from nuts and oils for saturated fat on inflammation in normal weight and obese individuals
Fasting glucose and HbA1C | 10 weeks
  Compare the effect of substitution of unsaturated fat from nuts and oils for saturated fat on fasting glucose and HbA1C

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo Universitetssykehus, Ullevål, Oslo, Norway

REFERENCES:
- [Derived] Sundfor TM, Svendsen M, Heggen E, Dushanov S, Klemsdal TO, Tonstad S. BMI modifies the effect of dietary fat on atherogenic lipids: a randomized clinical trial. Am J Clin Nutr. 2019 Oct 1;110(4):832-841. doi: 10.1093/ajcn/nqz113. PMID 31216575